CLINICAL TRIAL: NCT01734382
Title: A Phase IV Study to Evaluate Decreased Dose Frequency in Patients With Systemic Juvenile Arthritis (SJIA) Who Experience Laboratory Abnormalities During Treatment With Tocilizumab
Brief Title: A Study of Decreased Dose Frequency in Participants With Systemic Juvenile Arthritis Who Experience Laboratory Abnormalities During Treatment With RoActemra/Actemra (Tocilizumab)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WA28029; 2012-000444-10 (EudraCT Number)
Record Dates: First submitted 2012-11-22; First posted 2012-11-27 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Tocilizumab (TCZ) Q2W (Experimental): Participants will receive tocilizumab intravenous (IV) infusions (12 mg/kg for participants < 30 kg; 8 mg/kg for participants >/= 30 kg) once every other week (Q2W) up to 24 weeks or until occurrence of a protocol defined laboratory abnormality in Part 1 of the study.
  Interventions: Drug: Tocilizumab
- Part 2: TCZ IV 12 mg/kg Q3W/Q4W (Experimental): Participants with weight < 30 kg will receive tocilizumab IV infusions of 12 mg/kg once every three weeks (Q3W) up to 52 weeks or until occurrence of neutropenia, thrombocytopenia, or liver enzyme abnormality as per protocol criteria. Participants who complete 5 consecutive infusions of Q3W and have a laboratory abnormality of neutropenia, thrombocytopenia or elevated liver enzymes as per protocol criteria, after resolution of this laboratory abnormality will switch to tocilizumab IV infusions of 12 mg/kg once every four weeks (Q4W) up to Week 52 in Part 2 of the study.
  Interventions: Drug: Tocilizumab
- Part 2: TCZ IV 8 mg/kg Q3W/Q4W (Experimental): Participants with weight >/= 30 kg will receive tocilizumab IV infusions of 8 mg/kg Q3W up to 52 weeks or until occurrence of neutropenia, thrombocytopenia, or liver enzyme abnormality as per protocol criteria. Participants who complete 5 consecutive infusions of Q3W and have a laboratory abnormality of neutropenia, thrombocytopenia or elevated liver enzymes as per protocol criteria, after resolution of this laboratory abnormality will switch to tocilizumab IV infusions of 8 mg/kg Q4W up to Week 52 in Part 2 of the study.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Participants will receive tocilizumab IV infusions of 12 mg/kg (for participants < 30 kg) or 8 mg/kg (for participants >/=30 kg) Q2W/Q3W/Q4W.
  Other Names: RoActemra/Actemra

SUMMARY:
PART1 Participants in Part 1 (Run-in-Phase) of study will receive tocilizumab (TCZ) (RoActemra/Actemra) 12 milligrams per kilogram (mg/kg) or 8 mg/kg intravenously (IV) every 2 weeks (Q2W) for up to 24 weeks. Participants who experience a laboratory abnormality during Part 1 may be eligible to move into Part 2 of the study.

PART 2 This open-label Phase IV study will evaluate the efficacy, safety, pharmacokinetics, pharmacodynamics and immunogenicity of tocilizumab in reduced dose frequency in participants with adequately controlled systemic juvenile idiopathic arthritis who have experienced a laboratory abnormality on twice weekly tocilizumab dosing, that has since resolved. Participants will receive tocilizumab 12 mg/kg or 8 mg/kg intravenously every 3 weeks. After 5 consecutive infusions, participants who experience an event of neutropenia, thrombocytopenia or liver enzyme abnormality will move to every 4 weeks tocilizumab administration. Anticipated time on study treatment is 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

PART 1 and 2

* Children 2 to 17 years of age inclusive at screening
* Systemic juvenile idiopathic arthritis (sJIA) according to International League of Associations for Rheumatology (ILAR) classification (2001) and sJIA symptoms lasting for at least 1 month since diagnosis of sJIA
* Must meet one of the following:
* Not receiving methotrexate (MTX) or discontinued MTX at least 4 weeks prior to baseline visit, or
* Taking MTX for at least 12 weeks immediately prior to the baseline visit and on a stable dose of less than or equals (</=) 20 milligrams per meter square (mg/m^2) for at least 8 weeks prior to the baseline visit, together with either folic acid or folinic acid according to local standard of care
* Participants entering Part 1 who are naive to TCZ therapy must also meet the following inclusion criterion:
* History of inadequate clinical response (in the opinion of the treating physician) to Non steroidal Anti-Inflammatory Drugs (NSAIDs) and corticosteroids PART 2
* Juvenile Arthritis Disease Activity Score (JADAS) -71 score of 3.8 or less and absence of fever (related to sJIA) at screening and baseline
* Neutropenia, thrombocytopenia, or elevated Alanine transaminase/Aspartate transaminase (ALT/AST) previously experienced on the labeled dose (Q2W) of RoActemra/Actemra at any time
* Not currently receiving oral corticosteroids, or taking oral corticosteroids at a stable dose for a minimum of 2 weeks prior to baseline visit at no more than 10 milligrams per day (mg/day) or 0.2 miiligrams per kilogram per day (mg/kg/day), whichever is less
* Not taking (NSAIDs), or taking no more than 1 type of NSAID at a stable dose for a minimum of 2 weeks prior to the baseline visit, with the dose being less than or equal to the maximum recommended daily dose

Exclusion Criteria:

* Wheelchair bound or bedridden
* Any other auto-immune, rheumatic disease, or overlap syndrome other than sJIA
* Pregnant or lactating, or intending to become pregnant during study conduct and up to 6 months after the last administration of study drug
* Any significant concurrent medical or surgical condition which would jeopardize the participant's safety or ability to complete the trial
* History of significant allergic or infusion reactions to prior TCZ infusion, and/or presence of anti-TCZ antibodies at screening
* Inborn conditions characterized by a compromised immune system
* Known Human Immunodeficiency Virus (HIV) infection or other acquired forms of immune compromise
* History of alcohol, drug, or chemical abuse within 6 months of screening
* Evidence of serious uncontrolled concomitant diseases, including but not limited to the nervous, renal, hepatic, or endocrine systems
* Any active acute, subacute, chronic or recurrent bacterial, viral, or systemic fungal infection
* History of atypical tuberculosis (TB)
* Active TB requiring treatment within 2 years prior to the screening visit
* Positive purified protein derivative (PPD) at screening
* Any major episode of infection requiring hospitalization or treatment during screening or treatment with IV antibiotics completing within 4 weeks of the screening visit or oral antibiotics completing within 2 weeks of the screening visit
* History of reactivation or new onset of a systemic infection within 2 months of the screening visit
* Positive for hepatitis B or hepatitis C infection
* Chronic hepatitis, viral or pulmonary disease
* Significant cardiac or pulmonary disease
* History of or current cancer or lymphoma
* Uncontrolled diabetes mellitus
* History of or concurrent serious gastrointestinal disorders
* History of macrophage activation syndrome (MAS) within 3 months prior to screening visit

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2013-06-10 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- United States (2):
  - Children's Hospital Los Angeles; Division of Rheumatoogy, Los Angeles, California
  - Cincinnati Children'S Hospital Medical Center; Division of Rheumatology, Cincinnati, Ohio
- Argentina (2):
  - Hospital Gral de Niños Pedro Elizalde, Buenos Aires
  - Hospital Dr. Humberto Notti, Mendoza
- Alberta Children'S Hospital, Calgary, Alberta, Canada
- Germany (2):
  - Charité Campus; Virchow Klinikum Berlin, Berlin
  - Asklepios Klinik; Zentrum für Allgemeine Pädiatrie und Neonatologie, Sankt Augustin
- Israel (3):
  - Rambam Medicl Center, Ruth Children Hospital, Haifa
  - Meir Medical center, Pediatrics, Kfar Saba
  - Schneider Children's Medical Center of Israel, Petah Tikva
- Italy (2):
  - Irccs Ospedale Pediatrico Bambin Gesu - Dip. Di Medicina, Rome, Lazio
  - Univ. Di Padova - Dip. Di Pediatria - Unita' Reumatol. Pediatrica, Padua, Veneto
- Unidad de Reumatologia Rehabilitacion Integral; Centro Medico Del Angel, Mexicali, Mexico
- Russia (2):
  - SI Sceintific children health center RAMS, Moscow
  - Saint-Petersburg State; Pediatrics Medical Academy, Saint Petersburg
- Spain (3):
  - Hospital Sant Joan De Deu; Servicio de Reumatologia Pediatrica, Barcelona
  - Hospital Ramon y Cajal ; Servicio de Reumatologia, Madrid
  - Hospital de La Paz; Unidad de Reumatologia Pediatrica, Madrid
- Royal Liverpool Childrens Hospital; Rheumatology, Liverpool, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with systemic juvenile idiopathic arthritis (sJIA) were recruited at study sites in 8 countries. The study consisted of two parts: Part 1 was a 24-week Run-in period and Part 2 was a 52-week Main study.
Pre-assignment Details: Participants on tocilizumab (TCZ) once every two weeks (Q2W) who had experienced a laboratory abnormality (which resolved) as per protocol criteria either during Part 1 or prior to the study, could enter Part 2. 19 Participants entered Part 1 and 6 continued on to Part 2. 16 participants directly entered Part 2 of the study.
Groups:
- Part 1: Tocilizumab (TCZ) Q2W: Participants received tocilizumab intravenous (IV) infusions (12 mg/kg for participants < 30 kg; 8 mg/kg for participants >/= 30 kg) once every other week (Q2W) up to 24 weeks or until occurrence of a protocol defined laboratory abnormality in Part 1 of the study.
- Part 2: TCZ IV 12 mg/kg Q3W/Q4W: Participants with weight < 30 kg received tocilizumab IV infusions of 12 mg/kg once every three weeks (Q3W) up to 52 weeks or until occurrence of neutropenia, thrombocytopenia, or liver enzyme abnormality as per protocol criteria. Participants who completed 5 consecutive infusions of Q3W and had a laboratory abnormality of neutropenia, thrombocytopenia or elevated liver enzymes as per protocol criteria, after resolution of this laboratory abnormality switched to tocilizumab IV infusions of 12 mg/kg once every four weeks (Q4W) up to Week 52 in Part 2 of the study.
- Part 2: TCZ IV 8 mg/kg Q3W/Q4W: Participants with weight >/= 30 kg received tocilizumab IV infusions of 8 mg/kg Q3W up to 52 weeks or until occurrence of neutropenia, thrombocytopenia, or liver enzyme abnormality as per protocol criteria. Participants who completed 5 consecutive infusions of Q3W and had a laboratory abnormality of neutropenia, thrombocytopenia or elevated liver enzymes as per protocol criteria, after resolution of this laboratory abnormality switched to tocilizumab IV infusions of 8 mg/kg Q4W up to Week 52 in Part 2 of the study.
Period: Part 1
Arm/Group | Part 1: Tocilizumab (TCZ) Q2W | Part 2: TCZ IV 12 mg/kg Q3W/Q4W | Part 2: TCZ IV 8 mg/kg Q3W/Q4W
Started | 19 | 0 | 0
Completed | 17 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Period: Part 2
Arm/Group | Part 1: Tocilizumab (TCZ) Q2W | Part 2: TCZ IV 12 mg/kg Q3W/Q4W | Part 2: TCZ IV 8 mg/kg Q3W/Q4W
Started | 0 | 7 | 15
Completed | 0 | 5 | 8
Not Completed | 0 | 2 | 7
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Other | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 3
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Part 1 enrolled 19. Patients treated with TCZ Q2W either during Part 1 or prior to the study, who experienced laboratory abnormalities and which had resolved, were allowed to enroll into Part 2. Part 2 enrolled 22 with 6 from Part 1 and 16 directly enrolled into Part 2. Baseline Characteristics are presented separately for Part 1 and Part 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Tocilizumab (TCZ) Q2W | Part 2: TCZ IV 12 mg/kg Q3W/Q4W | Part 2: TCZ IV 8 mg/kg Q3W/Q4W | Total
Number analyzed (Participants) | 19 | 7 | 15 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] — Part 1 participants Population: Part 1 of the study had 19 enrolled participants.
  years
    number analyzed (Participants) | 19 | 0 | 0 | 19
    (all) | 8.5 (3.6) |  |  | 8.5 (3.6)
Age, Continuous [Mean (Standard Deviation); unit: years] — Part 2 participants Population: Part 2 of the study had 22 enrolled participants, 6 of whom had completed Part 1 and 16 directly enrolled into Part 2.
  years
    number analyzed (Participants) | 0 | 7 | 15 | 22
    (all) |  | 6.7 (1.8) | 11.7 (2.8) | 10.1 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Part 1 participants Population: Part 1 of the study had 19 enrolled participants.
  Participants
    number analyzed (Participants) | 19 | 0 | 0 | 19
    Female | 9 | 0 | 0 | 9
    Male | 10 | 0 | 0 | 10
Sex: Female, Male [Count of Participants; unit: Participants] — Part 2 participants Population: Part 2 of the study had 22 enrolled participants, 6 of whom had completed Part 1 and 16 directly enrolled into Part 2.
  Participants
    number analyzed (Participants) | 0 | 7 | 15 | 22
    Female | 0 | 4 | 10 | 14
    Male | 0 | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Part 1 participants Population: Part 1 of the study had 19 enrolled participants.
  Participants
    number analyzed (Participants) | 19 | 0 | 0 | 19
    Hispanic or Latino | 6 | 0 | 0 | 6
    Not Hispanic or Latino | 13 | 0 | 0 | 13
    Unknown or Not Reported | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Part 2 participants Population: Part 2 of the study had 22 enrolled participants, 6 of whom had completed Part 1 and 16 directly enrolled into Part 2.
  Participants
    number analyzed (Participants) | 0 | 7 | 15 | 22
    Hispanic or Latino | 0 | 2 | 4 | 6
    Not Hispanic or Latino | 0 | 5 | 10 | 15
    Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Part 1 participants Population: Part 1 of the study had 19 enrolled participants.
  Participants
    number analyzed (Participants) | 19 | 0 | 0 | 19
    American Indian or Alaska Native | 1 | 0 | 0 | 1
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0
    White | 17 | 0 | 0 | 17
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Part 2 participants Population: Part 2 of the study had 22 enrolled participants, 6 of whom had completed Part 1 and 16 directly enrolled into Part 2.
  Participants
    number analyzed (Participants) | 0 | 7 | 15 | 22
    American Indian or Alaska Native | 0 | 1 | 2 | 3
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0
    White | 0 | 6 | 12 | 18
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Juvenile Arthritis Disease Activity Score (JADAS-71)
Description: JADAS-71 has 4 components: Physician global assessment of disease activity on a visual analog scale (VAS) (range=0-10, left end of line=arthritis inactive, i.e., symptom-free and no arthritis symptoms; right end=arthritis very active), patient/parent global assessment of overall well-being on VAS (range=0-10, left end of line=very well, right end=very poor), normalized erythrocyte sedimentation rate (ESR) (range=0-10, If ESR is ≤20 mm/h, set to 0. If ≥120 mm/h, set to 10 mm/h. If > 20 mm/h and < 120 mm/h, apply formula: [ESR-20 mm/h]/10 mm/h), and a count of active arthritis (swelling present or pain present and limitation of motion) in 71 selected joints (range=0-71). JADAS-71 is sum of 4 component scores, range=0-101. A higher score=more arthritis disease activity. Data reported for up to Week 52 was collected in Part 2: Q3W arms: Baseline, Weeks 3,6,9,12,24,36,48 and 51; Q4W arms: Baseline, Weeks 0,4,8,12,24,36 and 40.
Time Frame: Part 2: Up to 52 weeks
Population: All TCZ population, all participants who have received at least one dose of study drug. Number analyzed is the number of participants with data available at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Part 2: TCZ IV 12 mg/kg Q3W: Participants received tocilizumab 12 mg/kg IV infusions Q3W up to 52 weeks or until occurrence of neutropenia, thrombocytopenia, or liver enzyme abnormality as per protocol criteria.
- Part 2: TCZ IV 8 mg/kg Q3W: Participants received tocilizumab 8 mg/kg IV infusions Q3W up to 52 weeks or until occurrence of neutropenia, thrombocytopenia, or liver enzyme abnormality as per protocol criteria.
- Part 2: TCZ IV 12 mg/kg Q4W: Participants who completed 5 consecutive infusions of Q3W and had a laboratory abnormality of neutropenia, thrombocytopenia or elevated liver enzymes as per protocol criteria, after resolution of this laboratory abnormality switched to tocilizumab IV infusions of 12 mg/kg Q4W up to Week 52 in Part 2 of the study.
- Part 2: TCZ IV 8 mg/kg Q4W: Participants who completed 5 consecutive infusions of Q3W and had a laboratory abnormality of neutropenia, thrombocytopenia or elevated liver enzymes as per protocol criteria, after resolution of this laboratory abnormality switched to tocilizumab IV infusions of 8 mg/kg Q4W up to Week 52 in Part 2 of the study.
Arm/Group | Part 2: TCZ IV 12 mg/kg Q3W | Part 2: TCZ IV 8 mg/kg Q3W | Part 2: TCZ IV 12 mg/kg Q4W | Part 2: TCZ IV 8 mg/kg Q4W
Number analyzed (Participants) | 7 | 15 | 1 | 6
score on a scale
  Baseline | 0.60 (0.839) | 0.21 (0.247) | 0.00 (NA) — SD was not estimable for 1 participant. | 0.35 (0.295)
  Week 0: number analyzed (Participants) | 0 | 0 | 1 | 6
  Week 0 |  |  | 0.00 (NA) — SD was not estimable for 1 participant. | 0.13 (0.242)
  Week 3: number analyzed (Participants) | 7 | 15 | 0 | 0
  Week 3 | 1.60 (2.474) | 0.61 (0.913) |  |
  Week 4: number analyzed (Participants) | 0 | 0 | 1 | 6
  Week 4 |  |  | 0.00 (NA) — SD was not estimable for 1 participant. | 0.17 (0.266)
  Week 6: number analyzed (Participants) | 7 | 15 | 0 | 0
  Week 6 | 0.54 (0.812) | 0.39 (0.498) |  |
  Week 8: number analyzed (Participants) | 0 | 0 | 1 | 6
  Week 8 |  |  | 0.00 (NA) — SD was not estimable for 1 participant. | 0.20 (0.490)
  Week 9: number analyzed (Participants) | 7 | 15 | 0 | 0
  Week 9 | 2.59 (5.402) | 0.33 (0.420) |  |
  Week 12: number analyzed (Participants) | 6 | 14 | 1 | 6
  Week 12 | 0.30 (0.600) | 0.84 (2.318) | 0.00 (NA) — SD was not estimable for 1 participant. | 0.13 (0.327)
  Week 24: number analyzed (Participants) | 5 | 6 | 1 | 5
  Week 24 | 0.42 (0.576) | 0.05 (0.084) | 0.00 (NA) — SD was not estimable for 1 participant. | 0.20 (0.346)
  Week 36: number analyzed (Participants) | 4 | 4 | 1 | 4
  Week 36 | 0.48 (0.950) | 0.08 (0.150) | 0.00 (NA) — SD was not estimable for 1 participant. | 0.00 (0.000)
  Week 40: number analyzed (Participants) | 0 | 0 | 0 | 4
  Week 40 |  |  |  | 0.00 (0.000)
  Week 48: number analyzed (Participants) | 4 | 3 | 0 | 0
  Week 48 | 0.00 (0.000) | 0.17 (0.289) |  |
  Week 51: number analyzed (Participants) | 4 | 3 | 0 | 0
  Week 51 | 0.00 (0.000) | 0.17 (0.208) |  |

2. Primary Outcome: Number of Participants With Juvenile Idiopathic Arthritis (JIA) Disease Flare as Determined by JIA Core Variables in Part 2 of the Study
Description: JIA flare was defined as any 3 of the 6 core outcome variables worsening by at least 30% relative to baseline visit of Part 2, with no more than 1 of the remaining variables improving by more than 30%. For the number of joints with active arthritis or the number of joints with limitation of motion a minimum worsening of at least 2 joints had to be present. If the physician global assessment (PGA) or the parent/patient global assessment were used a minimum worsening of at least 2 units on a scale from 0 to 10 had be present. For erythrocyte sedimentation rate (ESR), a worsening of at least 30% was not considered if within normal ranges. The 6 core outcome variables: PGA of disease activity, parent/patient global assessment of overall well-being, number of joints with active arthritis, number of joints with limitation of movement, ESR (measure of acute phase reaction) and functional ability determined by Childhood Health Assessment Questionnaire (CHAQ) Disability Index.
Time Frame: Part 2: Up to 52 weeks
Population: All TCZ population, all participants who have received at least one dose of study drug. Number of participants analyzed is the number of participants with data available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: TCZ IV 12 mg/kg Q3W | Part 2: TCZ IV 8 mg/kg Q3W | Part 2: TCZ IV 12 mg/kg Q4W | Part 2: TCZ IV 8 mg/kg Q4W
Number analyzed (Participants) | 7 | 15 | 1 | 6
Participants | 1 | 3 | 0 | 1

3. Primary Outcome: Number of Participants With Fever Attributable to Systemic Juvenile Idiopathic Arthritis (sJIA) in Part 2 of the Study
Description: Absence of fever at screening visit was defined as a temperature measurement < 38 degree centigrades (C). Presence of fever at each study visit was defined as a temperature measurement ≥ 38 C.
Time Frame: Part 2: Up to 52 weeks
Population: All TCZ population, all participants who have received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: TCZ IV 12 mg/kg Q3W | Part 2: TCZ IV 8 mg/kg Q3W | Part 2: TCZ IV 12 mg/kg Q4W | Part 2: TCZ IV 8 mg/kg Q4W
Number analyzed (Participants) | 7 | 15 | 1 | 6
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With at Least One Adverse Event
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Part 1 - Baseline up to 24 weeks plus 12 weeks of safety follow up; Part 2 - Baseline up to 52 weeks plus 12 weeks of safety follow up
Population: Safety population, all participants who have received at least one dose of study drug and who have at least one post-baseline assessment of safety.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Tocilizumab (TCZ) Q2W | Part 2: TCZ IV 12 mg/kg Q3W/Q4W | Part 2: TCZ IV 8 mg/kg Q3W/Q4W
Number analyzed (Participants) | 19 | 7 | 15
Participants | 16 | 7 | 14

5. Secondary Outcome: Serum Interleukin-6 (IL-6) Protein Concentration in Part 2 of the Study
Time Frame: Part 2: Q3W arms: Pre-dose at Baseline, Weeks 3, 6, 9, 12, 24, 36, 48 and 51; Q4W arms: Pre-dose at Baseline, Weeks 0, 4, 8, 12, 24, 36 and 40
Population: Pharmacodynamic (PD) population, all participants who have received at least one dose of study drug and who have at least one post-baseline assessment of PD. Number analyzed is the number of participants with data available at the given timepoint.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Part 2: TCZ IV 12 mg/kg Q3W | Part 2: TCZ IV 8 mg/kg Q3W | Part 2: TCZ IV 12 mg/kg Q4W | Part 2: TCZ IV 8 mg/kg Q4W
Number analyzed (Participants) | 7 | 15 | 1 | 6
pg/mL
  Baseline: number analyzed (Participants) | 5 | 14 | 1 | 6
  Baseline | 36.340 (19.2413) | 23.453 (12.1440) | 51.500 (NA) — SD was not estimable for 1 participant. | 25.415 (15.0174)
  Week 0: number analyzed (Participants) | 0 | 0 | 0 | 4
  Week 0 |  |  |  | 33.000 (23.3195)
  Week 3: number analyzed (Participants) | 6 | 11 | 0 | 0
  Week 3 | 61.617 (75.5724) | 22.727 (7.0321) |  |
  Week 4: number analyzed (Participants) | 0 | 0 | 1 | 5
  Week 4 |  |  | 13.700 (NA) — SD was not estimable for 1 participant. | 28.364 (24.8937)
  Week 6: number analyzed (Participants) | 6 | 13 | 0 | 0
  Week 6 | 46.698 (50.7148) | 82.995 (216.2854) |  |
  Week 8: number analyzed (Participants) | 0 | 0 | 1 | 5
  Week 8 |  |  | 14.300 (NA) — SD was not estimable for 1 participant. | 30.580 (22.0335)
  Week 9: number analyzed (Participants) | 5 | 11 | 0 | 0
  Week 9 | 45.231 (46.2539) | 47.582 (37.2259) |  |
  Week 12: number analyzed (Participants) | 4 | 12 | 1 | 5
  Week 12 | 84.100 (57.8972) | 71.867 (156.4710) | 11.600 (NA) — SD was not estimable for 1 participant. | 29.662 (26.0053)
  Week 24: number analyzed (Participants) | 3 | 5 | 1 | 3
  Week 24 | 79.200 (44.8853) | 23.420 (14.5520) | 45.000 (NA) — SD was not estimable for 1 participant. | 29.393 (19.2760)
  Week 36: number analyzed (Participants) | 3 | 4 | 1 | 2
  Week 36 | 67.467 (84.7317) | 30.025 (16.5470) | 14.100 (NA) — SD was not estimable for 1 participant. | 21.500 (15.8392)
  Week 40: number analyzed (Participants) | 0 | 0 | 0 | 2
  Week 40 |  |  |  | 22.820 (24.0133)
  Week 48: number analyzed (Participants) | 3 | 3 | 0 | 0
  Week 48 | 14.533 (1.4154) | 15.400 (10.0936) |  |
  Week 51: number analyzed (Participants) | 3 | 1 | 0 | 0
  Week 51 | 17.523 (9.2077) | 5.060 (NA) — SD was not estimable for 1 participant. |  |

6. Secondary Outcome: Soluble IL-6 Receptor (sIL-6R) Protein Concentration in Part 2 of the Study
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ngEq/mL
Arm/Group | Part 2: TCZ IV 12 mg/kg Q3W | Part 2: TCZ IV 8 mg/kg Q3W | Part 2: TCZ IV 12 mg/kg Q4W | Part 2: TCZ IV 8 mg/kg Q4W
Number analyzed (Participants) | 7 | 15 | 1 | 6
ngEq/mL
  Baseline: number analyzed (Participants) | 7 | 14 | 1 | 6
  Baseline | 621.04 (443.779) | 735.16 (310.983) | 447.00 (NA) — SD was not estimable for 1 participant. | 855.00 (325.572)
  Week 0: number analyzed (Participants) | 0 | 0 | 1 | 6
  Week 0 |  |  | 72.50 (NA) — SD was not estimable for 1 participant. | 722.83 (229.530)
  Week 3: number analyzed (Participants) | 7 | 14 | 0 | 0
  Week 3 | 632.43 (261.172) | 707.73 (291.228) |  |
  Week 4: number analyzed (Participants) | 0 | 0 | 1 | 6
  Week 4 |  |  | 379.00 (NA) — SD was not estimable for 1 participant. | 653.00 (143.386)
  Week 6: number analyzed (Participants) | 6 | 15 | 0 | 0
  Week 6 | 518.67 (272.217) | 721.73 (253.114) |  |
  Week 8: number analyzed (Participants) | 0 | 0 | 1 | 6
  Week 8 |  |  | 434.00 (NA) — SD was not estimable for 1 participant. | 628.50 (145.891)
  Week 9: number analyzed (Participants) | 6 | 13 | 0 | 0
  Week 9 | 596.58 (318.685) | 646.92 (174.932) |  |
  Week 12: number analyzed (Participants) | 5 | 12 | 1 | 6
  Week 12 | 656.80 (123.611) | 666.75 (144.510) | 411.00 (NA) — SD was not estimable for 1 participant. | 645.33 (106.952)
  Week 24: number analyzed (Participants) | 5 | 6 | 1 | 4
  Week 24 | 574.54 (347.127) | 554.33 (124.498) | 519.00 (NA) — SD was not estimable for 1 participant. | 546.25 (330.265)
  Week 36: number analyzed (Participants) | 4 | 4 | 1 | 4
  Week 36 | 492.50 (258.445) | 646.00 (198.499) | 439.00 (NA) — SD was not estimable for 1 participant. | 599.75 (122.200)
  Week 40: number analyzed (Participants) | 0 | 0 | 0 | 4
  Week 40 |  |  |  | 609.50 (115.613)
  Week 48: number analyzed (Participants) | 3 | 3 | 0 | 0
  Week 48 | 551.00 (91.000) | 391.00 (220.293) |  |
  Week 51: number analyzed (Participants) | 2 | 2 | 0 | 0
  Week 51 | 651.00 (135.765) | 517.00 (140.007) |  |

7. Secondary Outcome: C-reactive Protein (CRP) Concentration in Part 2 of the Study
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Part 2: TCZ IV 12 mg/kg Q3W | Part 2: TCZ IV 8 mg/kg Q3W | Part 2: TCZ IV 12 mg/kg Q4W | Part 2: TCZ IV 8 mg/kg Q4W
Number analyzed (Participants) | 7 | 15 | 1 | 6
mg/L
  Baseline | 4.844 (12.2832) | 2.309 (6.9847) | 0.200 (NA) — SD was not estimable for 1 participant. | 0.958 (1.8575)
  Week 0: number analyzed (Participants) | 0 | 0 | 1 | 4
  Week 0 |  |  | 0.610 (NA) — SD was not estimable for 1 participant. | 0.200 (0.0000)
  Week 3: number analyzed (Participants) | 7 | 13 | 1 | 2
  Week 3 | 0.223 (0.0427) | 0.216 (0.0407) | 0.200 (NA) — SD was not estimable for 1 participant. | 0.200 (0.0000)
  Week 4: number analyzed (Participants) | 0 | 0 | 1 | 6
  Week 4 |  |  | 0.200 (NA) — SD was not estimable for 1 participant. | 0.200 (0.0000)
  Week 6: number analyzed (Participants) | 7 | 14 | 0 | 0
  Week 6 | 0.291 (0.1499) | 0.526 (1.0163) |  |
  Week 8: number analyzed (Participants) | 0 | 0 | 1 | 5
  Week 8 |  |  | 0.200 (NA) — SD was not estimable for 1 participant. | 0.200 (0.0000)
  Week 9: number analyzed (Participants) | 5 | 11 | 1 | 3
  Week 9 | 0.208 (0.0179) | 0.255 (0.1250) | 0.200 (NA) — SD was not estimable for 1 participant. | 0.200 (0.0000)
  Week 12: number analyzed (Participants) | 5 | 11 | 1 | 6
  Week 12 | 0.200 (0.0000) | 0.238 (0.1201) | 0.200 (NA) — SD was not estimable for 1 participant. | 0.203 (0.0082)
  Week 24: number analyzed (Participants) | 5 | 5 | 1 | 5
  Week 24 | 0.280 (0.1789) | 0.254 (0.1207) | 0.200 (NA) — SD was not estimable for 1 participant. | 4.040 (8.5865)
  Week 36: number analyzed (Participants) | 4 | 4 | 1 | 4
  Week 36 | 0.225 (0.0500) | 0.200 (0.0000) | 0.200 (NA) — SD was not estimable for 1 participant. | 0.200 (0.0000)
  Week 40: number analyzed (Participants) | 0 | 0 | 0 | 4
  Week 40 |  |  |  | 0.200 (0.0000)
  Week 48: number analyzed (Participants) | 4 | 3 | 0 | 0
  Week 48 | 0.200 (0.0000) | 0.820 (1.0739) |  |
  Week 51: number analyzed (Participants) | 4 | 3 | 0 | 0
  Week 51 | 0.318 (0.2350) | 0.200 (0.0000) |  |

8. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR) in Part 2 of the Study
Time Frame: as for outcome 5
Population: PD population, all participants who have received at least one dose of study drug and who have at least one post-baseline assessment of PD. Number analyzed is the number of participants with data available at the given timepoint.
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | Part 2: TCZ IV 12 mg/kg Q3W | Part 2: TCZ IV 8 mg/kg Q3W | Part 2: TCZ IV 12 mg/kg Q4W | Part 2: TCZ IV 8 mg/kg Q4W
Number analyzed (Participants) | 7 | 15 | 1 | 6
mm/h
  Baseline | 3.43 (5.192) | 3.00 (1.852) | 1.00 (NA) — SD was not estimable for 1 participant. | 3.17 (1.602)
  Week 0: number analyzed (Participants) | 0 | 0 | 1 | 6
  Week 0 |  |  | 4.00 (NA) — SD was not estimable for 1 participant. | 2.67 (1.633)
  Week 3: number analyzed (Participants) | 7 | 14 | 1 | 4
  Week 3 | 2.86 (2.035) | 3.57 (2.709) | 2.00 (NA) — SD was not estimable for 1 participant. | 2.75 (0.957)
  Week 4: number analyzed (Participants) | 0 | 0 | 1 | 6
  Week 4 |  |  | 1.00 (NA) — SD was not estimable for 1 participant. | 3.17 (1.722)
  Week 6: number analyzed (Participants) | 7 | 15 | 0 | 0
  Week 6 | 4.14 (4.598) | 4.13 (3.681) |  |
  Week 8: number analyzed (Participants) | 0 | 0 | 1 | 6
  Week 8 |  |  | 1.00 (NA) — SD was not estimable for 1 participant. | 3.33 (2.160)
  Week 9: number analyzed (Participants) | 6 | 13 | 1 | 4
  Week 9 | 2.50 (2.510) | 3.23 (2.204) | 3.00 (NA) — SD was not estimable for 1 participant. | 2.25 (0.957)
  Week 12: number analyzed (Participants) | 5 | 12 | 1 | 6
  Week 12 | 2.20 (1.789) | 3.92 (3.315) | 1.00 (NA) — SD was not estimable for 1 participant. | 4.50 (3.209)
  Week 24: number analyzed (Participants) | 5 | 6 | 1 | 5
  Week 24 | 2.80 (1.304) | 3.17 (2.137) | 1.00 (NA) — SD was not estimable for 1 participant. | 2.80 (1.789)
  Week 36: number analyzed (Participants) | 4 | 4 | 1 | 4
  Week 36 | 2.25 (2.217) | 4.50 (2.646) | 1.00 (NA) — SD was not estimable for 1 participant. | 2.25 (1.893)
  Week 40: number analyzed (Participants) | 0 | 0 | 0 | 4
  Week 40 |  |  |  | 2.25 (1.893)
  Week 48: number analyzed (Participants) | 4 | 3 | 0 | 0
  Week 48 | 3.00 (0.816) | 4.67 (1.528) |  |
  Week 51: number analyzed (Participants) | 4 | 3 | 0 | 0
  Week 51 | 1.75 (1.708) | 6.00 (3.000) |  |

9. Secondary Outcome: Number of Participants With Anti-TCZ Antibodies in Part 2 of the Study
Time Frame: Part 2: Up to Week 52
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: TCZ IV 12 mg/kg Q3W | Part 2: TCZ IV 8 mg/kg Q3W | Part 2: TCZ IV 12 mg/kg Q4W | Part 2: TCZ IV 8 mg/kg Q4W
Number analyzed (Participants) | 7 | 15 | 1 | 6
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Serum TCZ Concentration in Part 2 of the Study
Time Frame: as for outcome 5
Population: All TCZ population in Part 2, all participants who have received at least one dose of study drug in Part 2. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Part 2: TCZ IV 12 mg/kg Q3W | Part 2: TCZ IV 8 mg/kg Q3W | Part 2: TCZ IV 12 mg/kg Q4W | Part 2: TCZ IV 8 mg/kg Q4W
Number analyzed (Participants) | 7 | 15 | 1 | 6
ug/mL
  Baseline: number analyzed (Participants) | 6 | 13 | 1 | 6
  Baseline | 29.916 (35.8002) | 44.210 (33.2547) | 9.520 (NA) — SD was not estimable for 1 participant. | 53.622 (48.5163)
  Week 0: number analyzed (Participants) | 0 | 0 | 0 | 6
  Week 0 |  |  |  | 24.212 (13.1659)
  Week 3: number analyzed (Participants) | 7 | 13 | 0 | 0
  Week 3 | 26.420 (21.1844) | 37.239 (21.8192) |  |
  Week 4: number analyzed (Participants) | 0 | 0 | 1 | 6
  Week 4 |  |  | 11.100 (NA) — SD was not estimable for 1 participant. | 17.718 (11.1580)
  Week 6: number analyzed (Participants) | 5 | 14 | 0 | 0
  Week 6 | 28.636 (13.5744) | 30.482 (19.2402) |  |
  Week 8: number analyzed (Participants) | 0 | 0 | 1 | 6
  Week 8 |  |  | 22.800 (NA) — SD was not estimable for 1 participant. | 17.578 (13.0611)
  Week 9: number analyzed (Participants) | 5 | 13 | 0 | 0
  Week 9 | 32.020 (6.3739) | 26.962 (17.9122) |  |
  Week 12: number analyzed (Participants) | 4 | 12 | 1 | 6
  Week 12 | 37.600 (20.5254) | 44.763 (77.1798) | 23.800 (NA) — SD was not estimable for 1 participant. | 15.442 (11.0714)
  Week 24: number analyzed (Participants) | 4 | 5 | 1 | 3
  Week 24 | 24.363 (20.3686) | 20.842 (25.9417) | 30.300 (NA) — SD was not estimable for 1 participant. | 16.030 (14.2124)
  Week 36: number analyzed (Participants) | 3 | 4 | 1 | 4
  Week 36 | 30.517 (18.6058) | 19.733 (8.2218) | 19.800 (NA) — SD was not estimable for 1 participant. | 12.903 (11.1808)
  Week 40: number analyzed (Participants) | 0 | 0 | 0 | 4
  Week 40 |  |  |  | 28.778 (16.0031)
  Week 48: number analyzed (Participants) | 3 | 2 | 0 | 0
  Week 48 | 25.433 (34.3053) | 22.950 (0.9192) |  |
  Week 51: number analyzed (Participants) | 3 | 2 | 0 | 0
  Week 51 | 12.207 (8.5862) | 10.945 (14.6449) |  |

11. Secondary Outcome: Baseline Childhood Health Assessment Questionnaire (CHAQ) Disability Index in Part 2 of the Study
Description: CHAQ- Disability Index consists of 30 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities-distributed, among a total of 30 items. Each question was rated on 4-point scale with range 0=no difficulty to 3=unable to do. To calculate overall score, participant must have a domain score in at least 6 of 8 domains. Scores were averaged to calculate CHAQ disability index, range is 0=no/minimal physical dysfunction)-3=very severe physical dysfunction, higher score indicates more disability.
Time Frame: Baseline of Part 2
Population: All TCZ population, all participants who have received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2: TCZ IV 12 mg/kg Q3W | Part 2: TCZ IV 8 mg/kg Q3W | Part 2: TCZ IV 12 mg/kg Q4W | Part 2: TCZ IV 8 mg/kg Q4W
Number analyzed (Participants) | 7 | 15 | 1 | 6
score on a scale | 0.0000 (0.00000) | 0.0417 (0.09047) | 0.0000 (NA) — SD was not estimable for 1 participant. | 0.0000 (0.00000)

12. Secondary Outcome: Change From Baseline in Childhood Health Assessment Questionnaire (CHAQ) Disability Index in Part 2 of the Study
Description: CHAQ- Disability Index consists of 30 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities-distributed, among a total of 30 items. Each question was rated on 4-point scale with range 0=no difficulty to 3=unable to do. To calculate overall score, participant must have a domain score in at least 6 of 8 domains. Scores were averaged to calculate CHAQ disability index, range is 0=no/minimal physical dysfunction)-3=very severe physical dysfunction, higher score indicates more disability. Negative change from baseline indicates an improvement.
Time Frame: Baseline; Part 2: Q3W arm groups - Weeks 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48 and 51; Q4W arm groups - Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36 and 40
Population: All TCZ population, all participants who have received at least one dose of study drug. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2: TCZ IV 12 mg/kg Q3W | Part 2: TCZ IV 8 mg/kg Q3W | Part 2: TCZ IV 12 mg/kg Q4W | Part 2: TCZ IV 8 mg/kg Q4W
Number analyzed (Participants) | 7 | 15 | 1 | 6
score on a scale
  Change from Baseline at Week 0: number analyzed (Participants) | 0 | 0 | 1 | 6
  Change from Baseline at Week 0 |  |  | 0.0000 (NA) — SD was not estimable for 1 participant. | 0.0000 (0.00000)
  Change from Baseline at Week 3: number analyzed (Participants) | 7 | 15 | 0 | 0
  Change from Baseline at Week 3 | 0.2500 (0.66144) | 0.0167 (0.25384) |  |
  Change from Baseline at Week 4: number analyzed (Participants) | 0 | 0 | 1 | 6
  Change from Baseline at Week 4 |  |  | 0.0000 (NA) — SD was not estimable for 1 participant. | 0.0000 (0.00000)
  Change from Baseline at Week 6: number analyzed (Participants) | 7 | 15 | 0 | 0
  Change from Baseline at Week 6 | 0.1071 (0.28347) | -0.0083 (0.07420) |  |
  Change from Baseline at Week 8: number analyzed (Participants) | 0 | 0 | 1 | 6
  Change from Baseline at Week 8 |  |  | 0.0000 (NA) — SD was not estimable for 1 participant. | 0.0000 (0.00000)
  Change from Baseline at Week 9: number analyzed (Participants) | 7 | 14 | 0 | 0
  Change from Baseline at Week 9 | 0.2500 (0.51539) | -0.0268 (0.10022) |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 5 | 13 | 1 | 6
  Change from Baseline at Week 12 | 0.1250 (0.27951) | -0.0481 (0.09599) | 0.0000 (NA) — SD was not estimable for 1 participant. | 0.0000 (0.00000)
  Change from Baseline at Week 15: number analyzed (Participants) | 6 | 12 | 0 | 0
  Change from Baseline at Week 15 | 0.1458 (0.35722) | 0.1771 (0.54994) |  |
  Change from Baseline at Week 16: number analyzed (Participants) | 0 | 0 | 1 | 6
  Change from Baseline at Week 16 |  |  | 0.0000 (NA) — SD was not estimable for 1 participant. | 0.0000 (0.00000)
  Change from Baseline at Week 18: number analyzed (Participants) | 5 | 9 | 0 | 0
  Change from Baseline at Week 18 | 0.1000 (0.22361) | 0.2500 (0.85009) |  |
  Change from Baseline at Week 20: number analyzed (Participants) | 0 | 0 | 1 | 5
  Change from Baseline at Week 20 |  |  | 0.0000 (NA) — SD was not estimable for 1 participant. | 0.0000 (0.00000)
  Change from Baseline at Week 21: number analyzed (Participants) | 4 | 8 | 0 | 0
  Change from Baseline at Week 21 | 0.0000 (0.00000) | 0.2656 (0.90740) |  |
  Change from Baseline at Week 24: number analyzed (Participants) | 5 | 5 | 1 | 5
  Change from Baseline at Week 24 | 0.1250 (0.27951) | -0.0750 (0.11180) | 0.0000 (NA) — SD was not estimable for 1 participant. | 0.0000 (0.00000)
  Change from Baseline at Week 27: number analyzed (Participants) | 4 | 4 | 0 | 0
  Change from Baseline at Week 27 | 0.0000 (0.00000) | 0.0000 (0.10206) |  |
  Change from Baseline at Week 28: number analyzed (Participants) | 0 | 0 | 1 | 5
  Change from Baseline at Week 28 |  |  | 0.0000 (NA) — SD was not estimable for 1 participant. | 0.0000 (0.00000)
  Change from Baseline at Week 30: number analyzed (Participants) | 4 | 3 | 0 | 0
  Change from Baseline at Week 30 | 0.0000 (0.00000) | 0.0000 (0.00000) |  |
  Change from Baseline at Week 32: number analyzed (Participants) | 0 | 0 | 1 | 5
  Change from Baseline at Week 32 |  |  | 0.0000 (NA) — SD was not estimable for 1 participant. | 0.0000 (0.00000)
  Change from Baseline at Week 33: number analyzed (Participants) | 4 | 3 | 0 | 0
  Change from Baseline at Week 33 | 0.0000 (0.00000) | -0.0417 (0.07217) |  |
  Change from Baseline at Week 36: number analyzed (Participants) | 4 | 3 | 1 | 4
  Change from Baseline at Week 36 | 0.0000 (0.00000) | 0.0417 (0.07217) | 0.0000 (NA) — SD was not estimable for 1 participant. | 0.0000 (0.00000)
  Change from Baseline at Week 39: number analyzed (Participants) | 4 | 3 | 0 | 0
  Change from Baseline at Week 39 | 0.0000 (0.00000) | -0.0417 (0.07217) |  |
  Change from Baseline at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 3
  Change from Baseline at Week 40 |  |  |  | 0.0000 (0.00000)
  Change from Baseline at Week 42: number analyzed (Participants) | 3 | 3 | 0 | 0
  Change from Baseline at Week 42 | 0.0000 (0.00000) | -0.0417 (0.07217) |  |
  Change from Baseline at Week 45: number analyzed (Participants) | 4 | 3 | 0 | 0
  Change from Baseline at Week 45 | 0.0000 (0.00000) | -0.0417 (0.07217) |  |
  Change from Baseline at Week 48: number analyzed (Participants) | 4 | 3 | 0 | 0
  Change from Baseline at Week 48 | 0.0000 (0.00000) | -0.0417 (0.07217) |  |
  Change from Baseline at Week 51: number analyzed (Participants) | 4 | 3 | 0 | 0
  Change from Baseline at Week 51 | 0.0000 (0.00000) | -0.0417 (0.07217) |  |

13. Secondary Outcome: Baseline Participant's/Parent's Global Assessment of Overall Well-being Score in Part 2 of the Study
Description: Participant's/parent's global assessment of overall well-being was determined on a VAS (range = 0-100, left end of the line = very well, i.e., symptom-free and no arthritis disease activity; right end = very poor, i.e., maximum arthritis disease activity).
Time Frame: Baseline of Part 2
Population: All TCZ population, all participants who have received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2: TCZ IV 12 mg/kg Q3W | Part 2: TCZ IV 8 mg/kg Q3W | Part 2: TCZ IV 12 mg/kg Q4W | Part 2: TCZ IV 8 mg/kg Q4W
Number analyzed (Participants) | 7 | 15 | 1 | 6
score on a scale | 2.3 (3.95) | 1.6 (2.29) | 0.0 (NA) — SD was not estimable for 1 participant. | 2.5 (3.21)

14. Secondary Outcome: Change From Baseline in Participant's/Parent's Global Assessment of Overall Well-being Score in Part 2 of the Study
Description: Participant's/Parent's global assessment of overall well-being was determined on a VAS (range = 0-100, left end of the line = very well, i.e., symptom-free and no arthritis disease activity; right end = very poor, i.e., maximum arthritis disease activity). Reported is the change from baseline in VAS score with a negative change from baseline indicating an improvement.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2: TCZ IV 12 mg/kg Q3W | Part 2: TCZ IV 8 mg/kg Q3W | Part 2: TCZ IV 12 mg/kg Q4W | Part 2: TCZ IV 8 mg/kg Q4W
Number analyzed (Participants) | 7 | 15 | 1 | 6
score on a scale
  Change from Baseline at Week 0: number analyzed (Participants) | 0 | 0 | 1 | 6
  Change from Baseline at Week 0 |  |  | 0.0000 (NA) — SD was not estimable for 1 participant. | -1.2 (1.60)
  Change from Baseline at Week 3: number analyzed (Participants) | 7 | 15 | 0 | 0
  Change from Baseline at Week 3 | -0.3 (2.36) | 2.0 (6.12) |  |
  Change from Baseline at Week 4: number analyzed (Participants) | 0 | 0 | 1 | 6
  Change from Baseline at Week 4 |  |  | 0.0000 (NA) — SD was not estimable for 1 participant. | -1.2 (1.26)
  Change from Baseline at Week 6: number analyzed (Participants) | 7 | 15 | 0 | 0
  Change from Baseline at Week 6 | -1.6 (3.51) | 2.2 (4.55) |  |
  Change from Baseline at Week 8: number analyzed (Participants) | 0 | 0 | 1 | 6
  Change from Baseline at Week 8 |  |  | 0.0 (NA) — SD was not estimable for 1 participant. | -0.5 (3.56)
  Change from Baseline at Week 9: number analyzed (Participants) | 7 | 14 | 0 | 0
  Change from Baseline at Week 9 | 8.4 (26.48) | 0.1 (2.62) |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 5 | 13 | 1 | 6
  Change from Baseline at Week 12 | -1.6 (3.58) | -0.7 (2.32) | 0.0 (NA) — SD was not estimable for 1 participant. | -1.2 (2.56)
  Change from Baseline at Week 15: number analyzed (Participants) | 6 | 12 | 0 | 0
  Change from Baseline at Week 15 | -1.5 (3.67) | 7.1 (29.34) |  |
  Change from Baseline at Week 16: number analyzed (Participants) | 0 | 0 | 1 | 6
  Change from Baseline at Week 16 |  |  | 0.0 (NA) — SD was not estimable for 1 participant. | -1.5 (1.97)
  Change from Baseline at Week 18: number analyzed (Participants) | 5 | 9 | 0 | 0
  Change from Baseline at Week 18 | -1.4 (3.71) | 6.9 (23.26) |  |
  Change from Baseline at Week 20: number analyzed (Participants) | 0 | 0 | 1 | 5
  Change from Baseline at Week 20 |  |  | 0.0 (NA) — SD was not estimable for 1 participant. | -1.6 (2.61)
  Change from Baseline at Week 21: number analyzed (Participants) | 4 | 8 | 0 | 0
  Change from Baseline at Week 21 | 0.0 (0.00) | 9.9 (30.02) |  |
  Change from Baseline at Week 24: number analyzed (Participants) | 5 | 5 | 1 | 5
  Change from Baseline at Week 24 | -1.8 (4.02) | -0.8 (2.17) | 0.0 (NA) — SD was not estimable for 1 participant. | -1.0 (2.00)
  Change from Baseline at Week 27: number analyzed (Participants) | 4 | 4 | 0 | 0
  Change from Baseline at Week 27 | 0.0 (0.00) | 0.3 (2.87) |  |
  Change from Baseline at Week 28: number analyzed (Participants) | 0 | 0 | 1 | 5
  Change from Baseline at Week 28 |  |  | 0.0 (NA) — SD was not estimable for 1 participant. | -1.2 (2.39)
  Change from Baseline at Week 30: number analyzed (Participants) | 4 | 3 | 0 | 0
  Change from Baseline at Week 30 | 0.0 (0.00) | -0.3 (2.52) |  |
  Change from Baseline at Week 32: number analyzed (Participants) | 0 | 0 | 1 | 5
  Change from Baseline at Week 32 |  |  | 0.0 (NA) — SD was not estimable for 1 participant. | 5.4 (14.35)
  Change from Baseline at Week 33: number analyzed (Participants) | 4 | 3 | 0 | 0
  Change from Baseline at Week 33 | 25.0 (50.00) | 0.0 (3.00) |  |
  Change from Baseline at Week 36: number analyzed (Participants) | 4 | 3 | 1 | 4
  Change from Baseline at Week 36 | 0.3 (0.50) | 0.0 (3.00) | 0.0 (NA) — SD was not estimable for 1 participant. | -2.0 (2.83)
  Change from Baseline at Week 39: number analyzed (Participants) | 4 | 3 | 0 | 0
  Change from Baseline at Week 39 | 0.3 (0.50) | -1.0 (1.73) |  |
  Change from Baseline at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 3
  Change from Baseline at Week 40 |  |  |  | -2.7 (3.06)
  Change from Baseline at Week 42: number analyzed (Participants) | 3 | 3 | 0 | 0
  Change from Baseline at Week 42 | 0.0 (0.00) | -0.7 (2.08) |  |
  Change from Baseline at Week 45: number analyzed (Participants) | 4 | 3 | 0 | 0
  Change from Baseline at Week 45 | 0.0 (0.00) | 0.3 (3.51) |  |
  Change from Baseline at Week 48: number analyzed (Participants) | 4 | 3 | 0 | 0
  Change from Baseline at Week 48 | 0.0 (0.00) | 0.7 (4.04) |  |
  Change from Baseline at Week 51: number analyzed (Participants) | 4 | 3 | 0 | 0
  Change from Baseline at Week 51 | 0.0 (0.00) | 0.3 (3.51) |  |

ADVERSE EVENTS:
Time Frame: Part 1 - Up to 24 weeks plus 12 weeks safety follow up; Part 2 - Up to 52 weeks plus 12 weeks safety follow up
Description: Safety population, all participants who received at least one dose of study drug and who had at least one post-baseline assessment of safety.
Arm/Group | Part 1: Tocilizumab (TCZ) Q2W | Part 2: TCZ IV 12 mg/kg Q3W/Q4W | Part 2: TCZ IV 8 mg/kg Q3W/Q4W
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/7 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/7 | 1/15
Other Adverse Events (participants affected / at risk) | 16/19 | 7/7 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Tocilizumab (TCZ) Q2W (N=19) | Part 2: TCZ IV 12 mg/kg Q3W/Q4W (N=7) | Part 2: TCZ IV 8 mg/kg Q3W/Q4W (N=15)
HYPERTRANSAMINASAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
HAEMOPHAGOCYTIC LYMPHOHISTIOCYTOSIS (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part 1: Tocilizumab (TCZ) Q2W (N=19) | Part 2: TCZ IV 12 mg/kg Q3W/Q4W (N=7) | Part 2: TCZ IV 8 mg/kg Q3W/Q4W (N=15)
***NO CODING AVAILABLE*** (General disorders) | 0 (0) | 0 (0) | 1 (1)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (7)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 3 (4)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
EAR SWELLING (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (2)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
CYSTITIS (Infections and infestations) | 1 (3) | 0 (0) | 1 (1)
EAR INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
ENTEROBIASIS (Infections and infestations) | 2 (2) | 1 (2) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
MYCOPLASMA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 1 (2) | 1 (1) | 3 (7)
PARONYCHIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
PHARYNGITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (3) | 1 (1) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
TONSILLITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (4) | 0 (0) | 3 (5)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 2 (3) | 2 (2)
VIRAL RASH (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 3 (4) | 2 (2) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
JOINT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SKIN ABRASION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 0 (0) | 2 (2)
COMPLEMENT FACTOR C4 DECREASED (Investigations) | 0 (0) | 1 (1) | 2 (2)
EOSINOPHIL COUNT INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1) | 1 (1) | 0 (0)
LIVER FUNCTION TEST INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
LYMPHOCYTE MORPHOLOGY ABNORMAL (Investigations) | 0 (0) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
STILL'S DISEASE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
FEAR OF INJECTION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
CATARRH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 2 (2)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
TONSILLAR HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
BLISTER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
RASH (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0)
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
CATARACT SUBCAPSULAR (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
EYE PAIN (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
ANAL FISSURE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0) | 0 (0)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 (1) | 0/0 (0) | 0/0 (0)
HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0/0 (0) | 0/0 (0)
ASYMPTOMATIC BACTERIURIA (Infections and infestations) | 1 (1) | 0/0 (0) | 0/0 (0)
FUNGAL SKIN INFECTION (Infections and infestations) | 1 (1) | 0/0 (0) | 0/0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (2) | 0/0 (0) | 0/0 (0)
IMPETIGO (Infections and infestations) | 1 (1) | 0/0 (0) | 0/0 (0)
OTITIS EXTERNA (Infections and infestations) | 1 (1) | 0/0 (0) | 0/0 (0)
OTITIS MEDIA (Infections and infestations) | 1 (1) | 0/0 (0) | 0/0 (0)
PNEUMONIA MYCOPLASMAL (Infections and infestations) | 1 (1) | 0/0 (0) | 0/0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0/0 (0) | 0/0 (0)
TONSILLITIS STREPTOCOCCAL (Infections and infestations) | 1 (1) | 0/0 (0) | 0/0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 0 (0) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 (1) | 0 (0) | 0 (0)
ROSEOLOVIRUS TEST POSITIVE (Investigations) | 1 (1) | 0 (0) | 0 (0)
VITAMIN D DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0)
PRURIGO (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT01734382/Prot_SAP_000.pdf